CLINICAL TRIAL: NCT00633165
Title: A Phase II, Multicenter Study to Explore the Efficacy and Safety of Brostallicin in Patients With Myxoid Liposarcoma With (12:16) Translocation
Brief Title: Brostallicin Clinical Trial for Myxoid Liposarcoma
Acronym: SMI-BRS-202
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Systems Medicine LLC (Industry)
Responsible Party: Mary Jo Schreifels/Clinical Project Manager, Cell Therapeutics, Inc. (Systems Medicine, L.L.C. is a wholly owned subsidiary of CTI)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMI-BRS-202
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Myxoid Liposarcoma
Keywords: sarcoma; myxoid liposarcoma
MeSH Terms: conditions — Liposarcoma, Myxoid; Sarcoma | interventions — brostallicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Brostallicin — Patients will receive Brostallicin administered intravenously (IV) over 10 minutes at a dose of 10 mg/m2 on day one of a 21-day cycle. Safety and efficacy will be closely monitored and assessed.

SUMMARY:
This is a Phase II, multicenter, open-label clinical trial designed to determine the efficacy and safety of Brostallicin when administered once every 3 weeks in patients with myxoid liposarcoma with (12;16) translocation. The primary objective of this study is to determine the response rate following Brostallicin administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided informed consent.
2. Histologically confirmed myxoid liposarcoma.
3. Patients with metastatic and/or unresectable myxoid liposarcoma that is progressive and standard curative measures do not exist or are no longer effective.
4. Patient has measurable tumor on CT, spiral CT, or MRI scan that meet RECIST criteria.
5. Age ≥18 years
6. Karnofsky performance status (KPS) ≥ 70% (see Appendix III).
7. Life expectancy of at least 3 months.
8. Acceptable liver function:

   * Bilirubin ≤ 1.5 times upper limit of normal (ULN)
   * AST (SGOT), ALT (SGPT) and alkaline phosphatase ≤ 2.5 times ULN (if liver metastases are present, then ≤ 5 × ULN is allowed).
9. Acceptable renal function: For all patients serum creatinine within normal limits, OR calculated creatinine clearance ≥ 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.
10. Acceptable hematologic status:

    * Absolute neutrophil count (ANC) ≥ 1500 cells/mm(3) (1.5 ×10(9)/L)
    * Platelet count ≥ 100,000 platelet/mm(3) (100 ×10(9)/L)
    * Hemoglobin ≥ 9 g/dL.

Exclusion Criteria:

1. Patient received any of the following within the specified time period prior to initiation of treatment in this study:

   * Chemotherapy, major surgery, significant traumatic injury, or irradiation, whether conventional or investigational within 28 days
   * Mitomycin-C or nitrosurea within 42 days.
   * ET-743 at any time (Stage 1 only).
2. Patients heavily pretreated with chemotherapy and radiation, defined as follows:

   * ≥ 12 cycles of an alkylating agent-containing regimen, or
   * > 2 cycles carboplatin, or
   * > 2 cycles mitomycin C, or
   * irradiation to 25% of bone marrow-containing areas, or
   * high-dose chemotherapy requiring hematopoietic stem-cell reinfusion.
3. Known hypersensitivity to any study drug component.
4. Uncontrolled brain metastases in the judgement of the Investigator.
5. Abnormal cardiac or cardiovascular function, or serious cardiac illness or medical condition in the previous 6 months including, but not confined to:

   * New York Heart Association (NYHA) grade 2 or higher congestive heart failure (CHF) or who has had angioplasty or placement of coronary stents within the previous 6 months
   * Myocardial infarction within the past 6 months
   * High-risk uncontrolled arrhythmias
   * Angina pectoris that requires antianginal medication
   * Has clinically significant valvular heart disease
   * Evidence of transmural infarction on ECG
   * Poorly controlled hypertension (e.g., blood pressure: systolic >180 mm Hg or diastolic >100 mm Hg).
6. Pregnant or lactating females. All patients (males and females) who are fertile must agree to use an effective barrier method of birth control (i.e., latex condom, diaphragm, cervical cap, etc) to avoid pregnancy.
7. Not recovered from acute toxicity of all previous therapy prior to enrollment.
8. History of prior malignancies within 3 years, except for basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast.
9. Any evidence of serious and/or unstable pre-existing medical, psychiatric, or other condition (including laboratory abnormalities) that could interfere with patient safety or obtaining informed consent.
10. Any active uncontrolled infection including AIDS, hepatitis B or C.
11. Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
To determine the overall response rate and response rate, as measured by RECIST criteria of myxoid liposarcoma with (12;16) translocation, to Brostallicin. | Tumor measurements after every 2 cycles and there is no limit to the number of cycles.

SECONDARY OUTCOMES:
To describe the safety profile of Brostallicin when administered every 3 weeks in this patient population. | Tumor measurements after every 2 cycles and there is no limit to the number of cycles.
Duration of response | Tumor measurements after every 2 cycles and there is no limit to the number of cycles.
To determine progression free survival. | Tumor measurements after every 2 cycles and there is no limit to the number of cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Singer, M.D., Study Chair — CTI BioPharma
Locations (1):
- Sarcoma Oncology Center, Santa Monica, California, United States

REFERENCES:
- See also: Study Sponsor — http://www.celltherapeutics.com/subsidiaries